CLINICAL TRIAL: NCT03266107
Title: A Prospective, Open-Label, Single-Arm Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain
Brief Title: Study of Basivertebral Nerve Ablation Treatment of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relievant Medsystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0007 and CIP 0008
Record Dates: First submitted 2017-08-16; First posted 2017-08-29 (Actual); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Chronic Low Back Pain
Keywords: Vertebrogenic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): BVN Ablation
  Interventions: Device: Intracept

INTERVENTIONS:
Device: Intracept — Radiofrequency ablation of the basivertebral nerve using the Intracept System

SUMMARY:
Prospective, single arm, open label, multi-center study to evaluated the effectiveness of intraosseous basivertebral nerve radiofrequency ablation using the Intracept System.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm study of patients diagnosed with vertebrogenic low back pain for a minimum of 6 months with conservative care. Participants will receive the Intracept System procedure to ablate the basivertebral nerve within the vertebral body. Treatment is performed on all vertebral bodies with Modic type 1 or type 2 changes on MRI from L3-S1.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature subjects at least 25 years of age
* Chronic low back pain for at least 6 months
* Failure to respond to at least 6 months of non-operative conservative management
* Oswestry Disability Index (ODI) at least 30 points
* Modic changes Type 1 or 2

Exclusion Criteria:

* Current or history of vertebral cancer or spinal metastasis
* History of a fragility fracture
* Any back pathology related to trauma, evidence of vertebral compression fracture or other spinal pathology that could affect assessment of response to back pain
* Disc extrusion or protrusion

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eeric Truumees, MD, Principal Investigator — Independent; Kevin Macadaeg, MD, Principal Investigator — Independent
Locations (2):
- United States (2):
  - Indiana Spine Group, Carmel, Indiana
  - Seton Spine and Scoliosis Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Results
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: At the completion of trial
Access Criteria: Written request to study sponsor
URL: http://relievant.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients for the study were drawn from current low back pain clinic populations, referrals, and patient self-referral at two investigative sites in the U.S. from February 2018 to February 2019. Consecutively identified patients were screened for medical history and review of MRI for Modic/endplate changes and any excluded pain sources.
Groups:
- Treatment: Intracept - Intraosseous radiofrequency ablation of the basivertebral nerve using the Intracept System
Period: Enrollment to Procedure
Arm/Group | Treatment
Started | 50
Completed | 47
Not Completed | 3
Not completed — Failure to Access Due to Hardened Bone | 1
Not completed — Study stopped prior to Procedure | 2
Period: 3-Month Follow-up Visit
Arm/Group | Treatment
Started | 47
Completed | 46
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: 12-Month Follow-up Visit
Arm/Group | Treatment
Started | 46
Completed | 45
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intracept treated population
Groups:
- Treatment: Intracept
  Intracept: Radiofrequency ablation of the basivertebral nerve using the Intracept System
Arm/Group | Treatment
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.47 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47
Baseline Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: Total score on a scale of 0 to 100] — The Oswestry Disability Index (ODI) is a validated questionnaire of low back pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.
  Total score on a scale of 0 to 100 | 47.13 (9.87)
Baseline Visual Analog Scale (VAS) for Low Back Pain [Mean (Standard Deviation); unit: Scale 0 to 10] — Visual Analog Scale (VAS) for low back pain is a patient-rated 10-point numeric scale with 0 being no pain and 10 being worst imaginable pain.
  Scale 0 to 10 | 6.82 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Disability Index (ODI) - 3 Months
Description: Change in mean Oswestry Disability Index (ODI) total score from baseline to 3 months post-treatment. ODI total score scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference in ODI from baseline is considered to be a 10 points reduction from baseline.
Time Frame: 3 months
Population: Basivertebral nerve ablation treated participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 46
units on a scale | -30.33 (12.71)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < 0.001, t-test, 1 sided

2. Secondary Outcome: Visual Analog Scale (VAS) - 3 Months
Description: Change in the mean visual analog scale (VAS) low back pain from baseline to 3 months post treatment. VAS is a 10 point numeric scale with 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference is a 2 point reduction from baseline.
Time Frame: 3 Months
Population: Basivertebral nerve ablation treated participants with a 3 month visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment: BVN Ablation Radiofrequency ablation of the basivertebral nerve using the Intracept System
Arm/Group | Treatment
Number analyzed (Participants) | 46
units on a scale | -3.79 (2.2)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < 0.001, t-test, 1 sided

3. Secondary Outcome: ODI Responder Rate - 3-Month
Description: Number & percent of patients with greater than or equal to 15 point reduction in Oswestry Disability Index (ODI) from baseline to 3 months post treatment. ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be 10 points.
Time Frame: 3 Months
Population: Basivertebral nerve ablation treated participants with a 3 month visit
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 46
Participants | 42

4. Secondary Outcome: VAS Responder Rate - 3 Month
Description: Number and percentage of participants with a greater than or equal to 2 point reduction from baseline in visual analog scale (VAS) for low back pain at 3 months post treatment. VAS is a patient-reported 10 point numeric pain scale with 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference in VAS from baseline is a 2 point reduction.
Time Frame: 3 Months
Population: Basivertebral nerve ablation treated participants with a 3 month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 46
Participants | 36

5. Secondary Outcome: ODI -12 Months
Description: Change in mean Oswestry Disability Index (ODI) total score from baseline to 12 months post treatment. ODI total score is on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be 10 point reduction in ODI.
Time Frame: 12 Months
Population: Basivertebral nerve ablation treated participants with a 12 month visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 45
units on a scale | -32.31 (14.07)
Statistical Analysis 1: Comparison: Treatment; Test type: Superiority; p < 0.001, t-test, 1 sided

6. Secondary Outcome: VAS - 12 Month
Description: Change in mean visual analog scale (VAS) for low back pain score from baseline at 12 months. VAS is a patient-reported 10 point numeric pain scale with 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference in VAS from baseline is a 2 point reduction.
Time Frame: 12 Months
Population: Basivertebral nerve ablation treated participants with 12-month follow-up visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 45
units on a scale | -4.31 (2.51)

7. Secondary Outcome: ODI Responder Rate - 12-Month
Description: Number and percent of patients with greater than or equal to 15 point reduction in Oswestry Disability Index (ODI) total score from baseline to 12 months post treatment. ODI total score scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference for this tool is considered to be 10 points.
Time Frame: 12 Months
Population: Basivertebral ablation treated participants with a 12 month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 45
Participants | 40

8. Secondary Outcome: VAS Responder Rate - 12 Months
Description: Number and percent of participants with a reduction of greater than or equal to 2 points of the visual analog scale (VAS) at 12 months post treatment. VAS is a patient-reported 10 point numeric pain scale with 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference in VAS from baseline is a 2 point reduction in score.
Time Frame: 12 Months
Population: Basivertebral nerve ablation treated participants with a 12 month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 45
Participants | 36

9. Secondary Outcome: VAS Reduction 50% or More - 12 Month
Description: Number and percent of participants that reported a 50% or greater reduction in Visual Analog Scale (VAS) from baseline to 12 months.
Time Frame: 12 Months
Population: Basivertebral nerve ablation treated participants with a 12 month follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 45
Participants | 31

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 2/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=47)
Radiculitis (Musculoskeletal and connective tissue disorders) | 2 (2) — Transient leg pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03266107/Prot_SAP_000.pdf